CLINICAL TRIAL: NCT06511492
Title: Longitudinal Surveillance of Rectal Colonization and Transmission by Resistant Bacteria in Acutely Decompensated Cirrhosis: a Cohort Study
Brief Title: Longitudinal Surveillance of Rectal Colonization and Transmission by Resistant Bacteria in Acutely Decompensated Cirrhosis
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-469
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Cirrhosis, Liver; Rectal Colonization; Multidrug Resistance Organisms
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention in this study — No intervention in this study

SUMMARY:
Antimicrobial resistance has emerged as a global threat, and multidrug resistance organisms (MDROs) form one of the foremost challenges in the setting of decompensated cirrhosis. In a worldwide study, a high prevalence (34%) of infection with MDR bacteria in patients with cirrhosis and associated with higher in-hospital mortality.

Previous study indicated that the pattern of colonized bacteria in heterogeneous and the colonization by MDROs is associated with increased risk of infection. Effort should be made to reduce the spread of MDR bacteria and improvement in prognosis in patents with cirrhosis. Currently, strategies suggested to prevent the spread of MDROs in cirrhosis, including rapid microbiological tests, new first-line antibiotic schedules, infection control practices and epidemiological surveillance.

Thus, for the aims of this cohort study are as following. Firstly, to characterize the burden, dynamics and risk factors associated with rectal colonization by MDROs in patients with cirrhosis. Secondly, to completely characterize the risk that asymptomatic carriers of MDROs, both to other patients and to themselves via collecting detailed longitudinal sampling and high-resolution typing. Lastly, to generate evidence for future policymaking for individualized antimicrobial decision rather than umbrella guidelines since the variance in the bacteriological profiles in different settings.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years old;
2. Inpatients;
3. Cirrhosis patients with acute decompensation;

Exclusion Criteria:

1. Patients decline any swab type;
2. Patients had liver resection or other organ transplantation;
3. Patients who had participated in, or are planning to participate in other clinical trial within the 3 months prior to enrollment;
4. Hospital stays <48 hours;
5. Not suitable to participate in this study judging by researchers;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis patients with acute decompensation
Sampling Method: Non-Probability Sample
Enrollment: 1289 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of rectal colonization by MDROs in patients with cirrhosis | 90 days
  The prevalence of rectal colonization by MDROs in patients with cirrhosis during hospitalization
The onset of infection with MDR bacteria in cirrhosis patients with asymptomatic carriers | 90 days
  The onset of infection with MDR bacteria in cirrhosis patients with asymptomatic carriers and describe the risk of colonization both to other patients and to themselves.

SECONDARY OUTCOMES:
The risk factors associated with rectal colonization by MDROs in patients with cirrhosis. | 90 days

IPD SHARING:
Plan to Share IPD: No